CLINICAL TRIAL: NCT00195572
Title: Post-Approved Phase III Study of 1-LV/5FU Therapy
Brief Title: Study Evaluating Isovorin in Advanced/Recurrent Gastric Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISO/5FU-10
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2009-08-13 (Estimated); Status verified 2009-08

CONDITIONS: Gastric Cancer
Keywords: Gastric Cancer; Advanced/Recurrent Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Leucovorin; titanium silicide

INTERVENTIONS:
Drug: Isovorin
Drug: TS-1

SUMMARY:
The purpose of the study is to verify non-inferiority of survival time between Isovorin/5-fluorouracil (1-LV/5FU) therapy and TS-1 therapy in patients with inoperable advanced or recurrent gastric cancer. Secondary endpoints include response rates, duration of responses, time to progression (TTP) safety and quality of life (QOL).

ELIGIBILITY:
Inclusion Criteria:

* Gastric cancer diagnosed histologically or cytologically
* Normal organ function of bone marrow, heart, liver and kidney
* Age of 20-77

Other inclusion applies

Exclusion Criteria:

* Serious infection, heart disease, complication or organ disorder
* Ongoing administration of flucytosine
* Pregnant or breastfeeding women

Other exclusion applies

Ages: 20 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2002-05; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Survival time

SECONDARY OUTCOMES:
Response rate, duration of response, time to progression, safety, quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (36):
- Japan (36):
  - Adachi-ku, Tokyo
  - Anjo
  - Aomori
  - Chiba
  - Chikushino-shi
  - Fukuoka
  - Fukuroi-shi
  - Funai-gun
  - Hiroshima
  - Ichihara-shi
  - Kanagawa
  - Kanazawa
  - Kisaradu-shi
  - Kitaadachi-gun
  - Koto-ku, Tokyo
  - Kyoto
  - Misawa-shi
  - Morioka
  - Nagasaki
  - Nagoya
  - Osaka
  - Ōmura
  - Saga
  - Sagamiharashi
  - Sapparo City
  - Sapporo
  - Sasebo-shi
  - Sendai
  - Shizuka
  - Shizuoka
  - Sizuoka-shi
  - Takatuki-si
  - Tsuchiura-shi
  - Tsukuba
  - Uji-shi
  - Yamagata